CLINICAL TRIAL: NCT01879644
Title: Neurofeedback Study ADHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NF-HC
Record Dates: First submitted 2013-05-28; First posted 2013-06-18 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: ADHD
Keywords: ADHD; Neurofeedback; Self-Management; Parental Psychoeducation; Social Support
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neurofeedback with Psychoeducation (NF + PE) (Active Comparator): Neurofeedback plus Parental Psychoeducation
  Interventions: Behavioral: NF; Behavioral: PE
- Self-Management with Psychoeducation (SM + PE) (Active Comparator): Self-management + parental psychoeducation
  Interventions: Behavioral: SM; Behavioral: PE
- NF+PE and additional Social Support (SU) (Active Comparator): Neurofeedback + parental psychoeducation enhanced with social support
  Interventions: Behavioral: NF; Behavioral: PE; Behavioral: SU
- SM+PE and additional Social Support (SU) (Active Comparator): Self-management + parental psychoeducation enhanced with social support
  Interventions: Behavioral: SM; Behavioral: PE; Behavioral: SU

INTERVENTIONS:
Behavioral: NF
  Arms: NF+PE and additional Social Support (SU); Neurofeedback with Psychoeducation (NF + PE)
Behavioral: SM
  Arms: SM+PE and additional Social Support (SU); Self-Management with Psychoeducation (SM + PE)
Behavioral: PE
Behavioral: SU
  Arms: NF+PE and additional Social Support (SU); SM+PE and additional Social Support (SU)

SUMMARY:
Neurofeedback has proved to be effective in treating Attention deficit hyperactivity disorder (ADHD) in experimental settings. This study investigates whether neurofeedback can be used as a therapeutic intervention in regular outpatient care. The investigators compare high frequent neurofeedback with high frequent self-management therapy and suppose that both result in comparable effects.

ELIGIBILITY:
Inclusion Criteria:

* children with ADHD aged 7 to 11
* full command of the German language.

Exclusion Criteria:

* IQ below 80

Children with symptoms of:

* inattention,
* hyperactivity or
* impulsivity due to other medical reasons such as:

  * hyperthyreosis,
  * autism,
  * epilepsy,
  * brain disorders and
  * any genetic or medical disorder associated with externalizing behavior that mimics ADHD.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Core ADHD symptoms (inattention/hyperactivity/impulsivity) objectively assessed with the computer based Qb-Test (go-no-go-task with infrared camera) | Pre-Post-Change-Design; change for core symptoms from baseline to after 12 weeks, 6 and 12 months
  Children perform the Qb-Test:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Conners Psychopathology Scores | Pre-Post-Change-Design; change from baseline to psychopathology scores after 12 weeks, 6 and 12 months
  Conners parents & teacher rating scales:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2

SECONDARY OUTCOMES:
Social Support | Pre-Post-Change-Design; change from baseline to social support scores after 12 weeks, 6 and 12 months
  Children's social support scale:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Self-Concept | Pre-Post-Change-Design; change from baseline to self-concept scores after 12 weeks, 6 and 12 months
  Children's self-concept interview:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Perceived Criticism | Pre-Post-Change-Design; change from baseline to perceived criticism scores after 12 weeks, 6 and 12 months
  Assessment of children's perceived criticism:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Parental Stress (ESF) | Pre-Post-Change-Design; change from baseline to parental stress scores after 12 weeks, 6 and 12 months
  Parent Stress Questionnaire:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Cortisol | Pre-Post-Change-Design; change from baseline to cortisol levels after 12 weeks, 6 and 12 month
  Assessed with hair-samples:
  * T1 baseline diagnostic before therapy, 1 week
  * T2 post assessment after 36 therapy sessions, expected average of 12 weeks
  * T3 catamnestic measurement 6 months after T2
  * T4 catamnestic measurement 12 months after T2
Blood/saliva samples for possible genetic correlates of therapy response | End of therapy after 36 sessions
  Either saliva sampling or blood samples for genotyping of ADHD candidate genes to establish possible correlates of therapy response

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps-University Marburg, Department of Psychology, Clinical Child and Adolescent Psychology, Marburg, Hesse, Germany

REFERENCES:
- [Result] Christiansen H, Reh V, Schmidt MH, Rief W. Slow cortical potential neurofeedback and self-management training in outpatient care for children with ADHD: study protocol and first preliminary results of a randomized controlled trial. Front Hum Neurosci. 2014 Nov 26;8:943. doi: 10.3389/fnhum.2014.00943. eCollection 2014. PMID 25505396
- [Derived] Korfmacher AK, Hirsch O, Chavanon ML, Albrecht B, Christiansen H. Self-management training vs. neurofeedback interventions for attention deficit hyperactivity disorder: Results of a randomized controlled treatment study. Front Psychiatry. 2022 Aug 18;13:969351. doi: 10.3389/fpsyt.2022.969351. eCollection 2022. PMID 36061275
- See also: Comparison of Neurofeedback and Self-Management Training in an outpatient clinic. — http://www.uni-marburg.de/fb04/ag-klin/downloads/adhsflyer.pdf